CLINICAL TRIAL: NCT06480058
Title: Determinants of Eating Disorder Risk in Pre-intervention Bariatric Surgery Candidates.
Brief Title: Predictors of Bariatric Surgery Weight Loss
Acronym: BariPredict
Status: Completed | Type: Observational
Sponsor: Kuwait University (Other)
Collaborators: Dasman Diabetes Institute (Other); Jaber Al Ahmad Al Sabah Hospital (Other)
Responsible Party: Principal Investigator, Dana AlTarrah, Assistant Professor, Kuwait University
Other Study IDs: 2023/2323; 2023/2323 (Other: Ministry of Health)
Record Dates: First submitted 2024-06-19; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Obesity, Mild; Obesity, Morbid; Diabete Mellitus; Diabetes Mellitus, Type 2; Eating Disorders
Keywords: Obesity; Metabolic disease; Eating disorder; Mental health
MeSH Terms: conditions — Obesity; Lymphoma, Follicular; Obesity, Morbid; Diabetes Mellitus; Diabetes Mellitus, Type 2; Feeding and Eating Disorders; Metabolic Diseases; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the observational cross-sectional study is to determine the prevalence and correlates of disordered eating among candidates for bariatric surgery in the BariPredict cohort.

The study aims to answer the following question on whether the prevalence of disordered eating is higher in individuals that are candidates of bariatric surgery compared to the general population with obesity.

DETAILED DESCRIPTION:
Participants referred to Jaber Al Ahmad Al Sabah Hospital, Hawalli, Kuwait, for bariatric surgery were consecutively screened for the study.

A cross-sectional analysis was performed on a subgroup of this cohort with complete baseline data. The analysis investigates the influence of psychological factors associated with obesity before bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Obesity BMI > 30 kg/m2
* 18 years and older

Exclusion Criteria:

* BMI < 30 kg/m2

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A cohort of patients attending a bariatric clinic
Sampling Method: Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Screening | 1 Day
  A validated SCOFF questionnaire will be self-administered to patients attending their first preoperative bariatric surgery appointment. The SCOFF questionnaire is a simple 5-question test developed to assess the possible presence of an eating disorder. The S in SCOFF stands for "sick" (to vomit). The O stands for "one stone" of weight (i.e., 6.35 kg). The letters C, F and F stand for "control", "fat" and "food" respectively. Although the SCOFF is not used for diagnostic purposes, a score of 2 or more positive answers raises the index of suspicion of eating disorders, highlighting the need for a more detailed psychological history .The SCOFF has been previously validated in Arab populations.

SECONDARY OUTCOMES:
Anxiety | 1 Day
  Kuwait University Anxiety Scale (KUAS)
  The Kuwait University Anxiety Scale will be used to measure level of anxiety. The 20-item scale will capture cognitive/affective anxiety (9 items), subjective anxiety or nervousness (7 items), and somatic anxiety (4 items) [4]. Responses use a 4-point Likert scale ranging from 1=rare, 2=sometimes, 3= often, 4= always to measure the level of anxiety . The cut offs to indicate anxiety include 0 - 21 normal, 22 - 42 mild anxiety, 42 - 63 moderate anxiety, 64 - 84 severe anxiety.
Depression | 1 Day
  Beck Inventory
  Psychological screening and assessment for anxiety and depression will be carried by a clinical psychologist using a validated questionnaire. The Beck Depression inventory which includes a 21-item multiple choice self-report inventory will be used to measure depressive symptoms within the last week. Each question includes a set of 4 possible choices of how a participant may feel. Choices are scored from 0 to 3, increasing in intensity. The cut-offs to indicate depression include 0 - 9 minimal depression, 10 - 18 mild depression, 19 - 29 moderate depression, 30 - 63 severe depression.
Obesity | 1 Day
  Height and weight will be measured using standard protocols by a qualified nurse during the patient's preoperative and post-operative appointments. Body Mass Index (BMI) will be calculated using WHO cut-off points to define obesity. Obese patients will be divided into different classes of obesity as the following: obese class I (BMI 30 - 34.9 kg/m2), obese class II (35 - 39.9 kg/m2) and obese class III (BMI > 40 kg/m2).

CONTACTS AND LOCATIONS:
Locations (1):
- Dana AlTarrah, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No